CLINICAL TRIAL: NCT05009576
Title: Comparative Study Using Negative Pressure Dressing With & Without Silver Alginate to Promote Healing in Chronic Wounds.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Mahak Ali, Principal investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: memonmehak
Record Dates: First submitted 2021-07-29; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Wound Healing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vac with silver (Active Comparator): wounds of patients will be covered with a vac dressing with single layer of Ag+ hydrocolloid dressings. Such pattern of dressing will be followed in every change of dressing in 48 hours.
  Interventions: Other: silver alginate
- simple VAC without silver alginate (Active Comparator): wounds of patients will be covered with VAC dressings only. Such pattern of dressing will be followed in every change of dressing in 48 hours.
  Interventions: Other: VAC dressing without silver alginate

INTERVENTIONS:
Other: silver alginate — silver alginate hydrofiber dressing
  Arms: vac with silver
Other: VAC dressing without silver alginate — vaccum assisted dressing
  Arms: simple VAC without silver alginate

SUMMARY:
The randomized control trial will be conducted in the Department of Plastic and Reconstructive Surgery at Dr. Ruth K.M. Pfau Civil Hospital Karachi.General population admitted in Civil Hospital Karachi, for wound coverage with skin grafting meetimg inclusion criteria will be included.

DETAILED DESCRIPTION:
Wound will be covered with negative pressure dressings that are composed of a sterile foam dressing surrounded by an occlusive film that adheres to the nearby, normal skin. Suction is applied to the dressing and a draining tube connect to a wall fixed assisted vacuum canister.

Patients will be provided with paper chits with A or B marked on it. Patients picking up A chit will be dealt as A group where wound will be covered with VAC dressings only where by patients picking up B chit will be dealt as B group where wound will be covered with a single layer of Ag+ hydrocolloid dressings. Such pattern of dressing will be followed in every change of dressing in 48 hours. The wound site will be photographed after every change of dressings. The wound site will be photographically monitored by a team of plastic surgeons to assess granulation tissue, by noting the size of wound, color and shine of granulation tissue and edema.

ELIGIBILITY:
Inclusion Criteria:

* Both genders above 18 years
* Wounds for more than 6 weeks
* History of trauma, tumor, congenital physical abnormalities
* Hemoglobin levels more than 10 g/dl
* Platelet count above 150 x 10E9/L
* Size of wound > 10*10cm.

Exclusion Criteria:

* Pressure ulcers
* Co-morbidities like diabetes or hypertension
* Bleeding vessels
* Presence of Necrotic tissue
* Malignancy in wounds

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2021-07-17 (Actual); Study Completion 2021-07-17 (Actual)

PRIMARY OUTCOMES:
Granulation tissue | 6 days
  The wound site will be photographically monitored by a team of plastic surgeons to assess granulation tissue, by noting the size of wound, color and shine of granulation tissue and edema and also by questionnare fillled by patient.
size of wound. | 6 days
  he wound site will be photographically monitored by a team of plastic surgeons to assess granulation tissue, by noting the size of wound, color and shine of granulation tissue and edema and also by questionnare fillled by patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Mahak, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No